CLINICAL TRIAL: NCT05008536
Title: Phase I Study to Evaluate the Safety and Effectiveness of Anti-BCMA CAR-NK Therapy in Relapsed or Refractory Multiple Myeloma
Brief Title: Anti-BCMA CAR-NK Cell Therapy for the Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xi Zhang, MD, Chef of Hematology Department, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCMA NK for MM
Record Dates: First submitted 2021-08-14; First posted 2021-08-17 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Anti-BCMA CAR-NK Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-BCMA CAR-NK Cells (Experimental): After preconditioning with chemotherapy, the Anti-BCMA CAR-NK Cells will be evaluated
  Interventions: Biological: Anti-BCMA CAR-NK Cells; Drug: Fludarabine; Drug: Cytoxan

INTERVENTIONS:
Biological: Anti-BCMA CAR-NK Cells — 1-3×10^6 /KG, 3-6×10^6 /KG, 0.6-1.2×10^7/KG Treatment follows a lymphodepletion
Drug: Fludarabine — recommendation: 30mg/m2 (D-5~D-3),determined by tumor burden at baseline.
Drug: Cytoxan — recommendation: 300-500mg/m2 (D-5~D-3),determined by tumor burden at baseline.

SUMMARY:
The purpose of this study is to infuse BCMA CAR-NK cells（Umbilical & Cord Blood (CB) Derived CAR-Engineered NK Cells） to the patients with relapsed and refractory multiple myeloma (MM), to assess the safety and feasibility of this strategy. The CAR enables the NK cells to recognize and kill the MM cells by targeting of BCMA, a protein expressed of the surface of the malignant plasma cells in MM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. According to the international standard for multiple myeloma，have information on medical examination proving the diagnosis of multiple myeloma.
3. Received at least 2 prior lines of treatment, including proteasome inhibitor and immunomodulator, no efficacy more than PD; disease progression or relapsed after disease remission and refractory or no remission after treated in the last time.
4. Measurable disease at screening as defined by any of the following: Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level veing as defined ；or light chain MM without measurable disease in the serum or the urine；serum immunoglobulin free light chain isease dL and abnormal serum immunoglobulin kappa/lambda free light chain ratio ；
5. ECOG Scores: 0~2（See Annex 3），the estimated survival time was more than 3 months;
6. During the screening period, the clinical laboratory values met the following criteria： Hemoglobins70g/L (did not receive red blood cell transfusion ≤7 days prior to laboratory tests，recombinant human erythropoietin is allowed); Platelet count >50×10^9/L (did not receive blood transfusion ≤7 days prior to laboratory tests); Neutrophil absolute count oietin is (did not receive supportive treatment lowed); Platelet count >50×10^9/L，allowed to use over growth factor support); ALT and AST ≤3×ULN；Total bilirubin ≤2.0× UNL；Creatinine clearance×40mL/min；corrected serum calcium L/minctordL (3.1 mmol/L), or free calcium ion or freedL(L( ommol/L); Prothrombin time and activated partial thromboplastin time ≤1.5×ULN.
7. The urine pregnancy test of female subjects of childbearing age should be negative and not in lactation;
8. Females of childbearing potential and males must use efficient contraception（form signing the ICF to the end of the trial）

Exclusion Criteria:

1. Have received CAR-NK therapy；
2. Have a history of allergy to any component of cell products;
3. Previous history of other malignancy;
4. Any unstable cardiovascular disease happened the informed consent form by themselves or their legal guardian;boratory tests); be infused using the "3 + 3" dos grade), severe arrhythmia that require drug interference, cardiac angioplasty/coronary stent implantation/cardiac bypass surgery ≤6 months prior to enrollment;
5. Have received allogeneic hematopoietic stem cell transplantation in 3 months for the treatment of multiple myeloma;
6. who has suffered from brain injury, consciousness disorder, epilepsy, more serious cerebral ischemia or cerebral hemorrhage disease;
7. There were live vaccinations within 4 weeks before admission;
8. Active hepatitis (positive for HBVDNA or HCVRNA), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to those with HIV infection;
9. Oxygen is needed to maintain adequate oxygen saturation;
10. Contraindications for fludarabine or cyclophosphamide treatment.
11. There was uncontrolled active infection;Patients with autoimmune diseases, immunodeficiency or other diseases requiring immunosuppressive （excluding glucocorticoid）therapy;
12. Pregnant or breasting-feeding women;
13. Subjects had a history of alcohol, drug or mental illness;
14. Any other condition that researcher think it is inappropriate for the subject to anticipate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR) | 2 monthes after infusion
  Response assessment per International Myeloma Working Group (IMWG) criteria
Incidence of dose limiting toxicity (DLTs) | within 2 monthes after infusion
  To characterize the safety, tolerability of Anti-BCMA CAR-NK Cells

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Response assessment per International Myeloma Working Group (IMWG) criteria
Duration of Response (DOR) | up to 24 months
  Response assessment per International Myeloma Working Group (IMWG) criteria

CONTACTS AND LOCATIONS:
Overall Officials: xi zhang, PhD/MD, Principal Investigator — Department of Hematology, Xinqiao Hospital
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No